CLINICAL TRIAL: NCT00663546
Title: Studies of P. Vivax and P. Falciparum Malaria in Cambodia
Brief Title: Malaria Studies in Cambodia
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908094; 08-I-N094
Record Dates: First submitted 2008-04-19; First posted 2008-04-22 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2013-12-05

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium; Hemoglobin E; Alpha-thalssemia; G6PD Deficiency
MeSH Terms: conditions — Malaria; Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study, conducted by the National Center for Parasitology, Entomology and Malaria Control of Cambodia s Ministry of Health and the National Institute of Allergy and Infectious Diseases, will explore whether the following factors confer protection against malaria and associated anemia: certain blood groups, the hemoglobin E variant, G6PD-deficiency and alpha-thalassemia. Malaria is caused by parasites (P. falciparum and P. vivax) that are transmitted to humans through mosquito bites. This protocol includes two studies, a cohort study and a P. vivax collection study.

Individuals are eligible for enrollment in the studies as follows:

Cohort study:

Residents of all ages of Kandal, Ekapheap and Sangkumthmey villages (Thmar Da commune) who plan to remain in Thmar Da commune for the next 5 years.

P. vivax collection study:

2 years of age and older

Participating in NIAID protocol 05-I- N210 ( Severe Malaria and Anti-malarial Drug Resistance in Cambodia ) and diagnosed with P. vivax malaria

Participants undergo the following procedures:

Cohort study:

Baseline evaluation, including the following:

* Collection of demographic information
* Malaria history, temperature measurement and review of current symptoms, if any
* Blood draw of 300 microliters
* Additional blood draw of 10 milliliters in selected adults 18 years of age and older

Treatment with artesunate-piperaquine at a commune health post for subjects who develop malaria

Contact once a year for 5 years to determine continued residency in Thmar Da commune

P. vivax collection study:

* Medical history and physical examination
* Hemoglobin level measurement
* Blood draw
* Treatment with chloroquine
* Blood draw 3 to 5 weeks after treatment in some patients 18 years of age or older

DETAILED DESCRIPTION:
Cohort study. Hemoglobin (Hb) and red blood cell (RBC) polymorphisms that give rise to HbE, alpha-thalassemia, G6PD-deficiency, and ABO blood groups occur at high frequency along the Thailand-Cambodia border, where Plasmodium vivax and P. falciparum have been and continue to be transmitted. To determine whether these Hb/RBC polymorphisms have been naturally selected because they confer protection against malaria and malaria-associated anemia, we will conduct a cohort study of ethnic Khmer in Cambodia. Approximately 1000 individuals of all ages will be genotyped for the four polymorphisms listed above and then followed for 5 years to determine the mean incidence rates for both P. vivax and P. falciparum malaria, stratified by genotype. Incidence rate ratios (IRRs) will be calculated for each polymorphism relative to the wildtype genotype. Differences between Hb levels during acute episodes of malaria and Hb levels at baseline will also be calculated to determine if Hb/RBC polymorphisms influence the degree of malaria-associated anemia.

P. vivax collection study. Unlike P. falciparum, P. vivax cannot be efficiently cultivated in vitro. Improved cultivation methods are needed to make progress on nearly all aspects of P. vivax malariology, including pathogenesis, naturally-acquired immunity, vaccination, and antimalarial drug resistance. We plan to improve both short- and long-term cultivation methods in order to test various hypotheses of P. vivax pathogenesis and protection. Using freshly obtained parasite isolates from individuals with P. vivax malaria, we will test whether Hb/RBC polymorphisms influence potentially pathogenic properties of P. vivax parasites, such as their ability to bind non-infected RBCs and other host cells. It is believed that P. vivax selectively invades reticutocytes. This tropism has frustrated attempts at long-term cultivation of this parasite, which requires a constant source of reticulocyte-rich blood not easily obtained even in developed countries. The host reticulocyte receptor that mediates the highly selective tropism of P. vivax has not been identified. Fresh P. vivax parasites will also be used in in vitro experiments to identify the putative receptor that defines reticulocyte tropism. Any P. vivax ligand that bound selectively to a reticulocyte receptor will then be discovered and worked up as a promising vaccine candidate.

ELIGIBILITY:
* INCLUSION CRITERIA: (Cohort Study)

Resident of Kandal, Ekapheap, and Sangkumthmey villages (Thmar Da commune), and no plans to leave the Thmar Da commune for the next 5 years.

Willingness to participate in the study as evidenced by informed consent of subjects or his/her parent or guardian, and willingness to come to commune health posts if he/she develops fever or other symptoms of malaria.

Individuals of all ages will be enrolled.

EXCLUSION CRITERIA: (Cohort Study)

Any condition that in the opinion of the investigator would render the subject unable to comply with the protocol (e.g., psychiatric disease).

Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected or to have AIDS).

INCLUSION CRITERIA: (P. vivax Collection Study)

P. vivax malaria (mono-infection).

Willingness to participate in the study as evidenced by informed consent of subjects or his/her parent or guardian.

Age greater than or equal to 2.

Hematocrit greater than or equal to 25%.

EXCLUSION CRITERIA: (P. vivax Collection Study)

Any condition that in the opinion of the investigator would render the subject unable to comply with the protocol (e.g., psychiatric disease).

Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected or to have AIDS).

Pregnancy.

Prior use of antimalarials during the past 2 months.

INCLUSION CRITERIA: (Cord and Peripheral Blood Collection Study)

Healthy male or female adults greater than or equal to 18 years old or healthy pregnant female adults greater than or equal to 18 years old.

Willingness to participate in the study as evidenced by informed consent.

EXCLUSION CRITERIA: (Cord and Peripheral Blood Collection Study)

Any condition that in the opinion of the investigator would render the subject unable to comply with the protocol (e.g., psychiatric disease).

Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected or to have AIDS).

INCLUSION CRITERIA: (Collection of peripheral blood for identifying and isolating memory B cells)

Healthy male or non- pregnant female adults greater than or equal to 18 years old.

Previous enrollment on the P. vivax collection study.

Willingness to participate in the study as evidenced by written informed consent.

EXCLUSION CRITERIA: (Collection of peripheral blood for identifying and isolating memory B cells)

For the follow-up blood draw (250 mL), symptomatic parasitemia with any species of Plasmodium.

For the follow-up blood draw (250 mL), hemoglobin level <9 g/dL.

For the follow-up blood draw (250 mL), weight <45 kg.

Any condition that in the opinion of the investigator would render the subject unable to comply with the protocol (e.g., psychiatric illness).

Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected or to have AIDS).

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1978 (Actual)
Dates: Start 2008-03-24; Study Completion 2013-12-05

CONTACTS AND LOCATIONS:
Overall Officials: Rick M Fairhurst, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- Cambodia (3):
  - National Center for Parasitology, Entomology, and Malaria Controk, Ministry of H, Phnom Penh
  - Preah Vihear Referral Hospital, Preah Vihear Province
  - Ratanakiri Referral Hospital, Ratanakiri Province

REFERENCES:
- [Background] Frischer H, Bowman J. Hemoglobin E, an oxidatively unstable mutation. J Lab Clin Med. 1975 Apr;85(4):531-9. PMID 1120926
- [Background] Lachant NA, Tanaka KR. Impaired antioxidant defense in hemoglobin E-containing erythrocytes: a mechanism protective against malaria? Am J Hematol. 1987 Nov;26(3):211-9. doi: 10.1002/ajh.2830260302. PMID 3674003
- [Background] Hill AV. Molecular epidemiology of the thalassaemias (including haemoglobin E). Baillieres Clin Haematol. 1992 Jan;5(1):209-38. doi: 10.1016/s0950-3536(11)80042-9. PMID 1596592
- [Derived] Fantin RF, Coelho CH, Berhe AD, Magalhaes LMD, Pereira DB, Salinas ND, Tolia NH, Amaratunga C, Suon S, Sagara I, Narum DL, Fujiwara RT, Abejon C, Campos-Neto A, Duffy PE, Bueno LL. Immunological characterization of a VIR protein family member (VIR-14) in Plasmodium vivax-infected subjects from different epidemiological regions in Africa and South America. PLoS Negl Trop Dis. 2023 Apr 7;17(4):e0011229. doi: 10.1371/journal.pntd.0011229. eCollection 2023 Apr. PMID 37027391
- [Derived] Hostetler JB, Sharma S, Bartholdson SJ, Wright GJ, Fairhurst RM, Rayner JC. A Library of Plasmodium vivax Recombinant Merozoite Proteins Reveals New Vaccine Candidates and Protein-Protein Interactions. PLoS Negl Trop Dis. 2015 Dec 23;9(12):e0004264. doi: 10.1371/journal.pntd.0004264. eCollection 2015 Dec. PMID 26701602
- [Derived] Amaratunga C, Sreng S, Mao S, Tullo GS, Anderson JM, Chuor CM, Suon S, Fairhurst RM. Chloroquine remains effective for treating Plasmodium vivax malaria in Pursat province, Western Cambodia. Antimicrob Agents Chemother. 2014 Oct;58(10):6270-2. doi: 10.1128/AAC.03026-14. Epub 2014 Jul 21. PMID 25049249